CLINICAL TRIAL: NCT06483672
Title: Furmonertinib Combined With Anlotinib in Lung Adenocarcinoma Patients With EGFR Mutations and Brain Metastases, a Prospective Phase II Single-arm Clinical Study
Brief Title: Furmonertinib Combined With Anlotinib in Lung Adenocarcinoma Patients With EGFR Mutations and Brain Metastases
Acronym: LungBrain001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/469-4212
Record Dates: First submitted 2024-05-23; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Adenocarcinoma of Lung Metastatic to Brain
Keywords: Adenocarcinoma of Lung; Brain metastasis; EGFR mutation
MeSH Terms: conditions — Adenocarcinoma of Lung; Brain Neoplasms | interventions — aflutinib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib combine with anlotinib (Experimental): Furmonertinib 80mg, once daily, orally Anlotinib 12mg, once daily (days 1-14, 21 days per cycle), orally
  Interventions: Drug: Furmonertinib; Drug: Anlotinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 80mg, once daily, orally
  Other Names: AST2818
Drug: Anlotinib — Anlotinib 12mg, once daily (days 1-14, 21 days per cycle), orally
  Other Names: No other intervention names

SUMMARY:
The goal of this clinical trial is to learn if furmonertinib plus anlotinib works to treat participants with lung adenocarcinoma with EGFR mutations and brain metastases. It will also learn about the safety of furmonertinib plus anlotinib. The main questions it aims to answer are:

* Does furmonertinib plus anlotinib increase the number of participants who has a significant tumor shrinkage?
* What medical problems do participants have when taking furmonertinib plus anlotinib? Researchers will evaluate the safety and efficacy of furmonertinib plus anlotinib.

Participants will:

* Take furmonertinib(every day) and anlotinib(two weeks on and one week off)
* Visit the clinic once every 3 weeks for checkups and tests.
* Keep a diary of their symptoms.

DETAILED DESCRIPTION:
The objective of this study is to explore the effectiveness and safety of furmonertinib and anlotinib as first-line treatment for patients with EGFR mutation and brain metastasis lung adenocarcinoma.

This clinical trial adopts a single-center, prospective, single-arm phase II trial design. Each 3 weeks constitute a treatment cycle until disease progression or intolerance.

After screening, eligible patients will be enrolled in the study. They will receive furmonertinib and anlotinib as first-line treatment. The patients will undergo regular visits, and researchers will collect data on efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged ≥18 years old;
* Histologically or cytopathologically confirmed non-small cell lung cancer (NSCLC) ;
* According to RANO-BM, the subject has at least 1 intracranial measurable lesion;
* Tumor tissue samples or blood samples are confirmed to be EGFR mutations;
* ECOG PS 0-1;
* Life expectancy >12 weeks;
* No prior systemic antitumor therapy for metastatic NSCLC

Exclusion Criteria:

* Patients without lung adenocarcinoma, including lung squamous cell carcinoma or mixed histological type, etc;
* Expected to receive other anti-tumor therapy other than the investigational product during the study;
* Having previously received systematic anti-tumor therapy
* Having received the following therapies: (1) Having been irradiated for > 30% bone marrow or a large area within 4 weeks prior to the first dose of investigational product; (2) Having received major surgery within 4 weeks prior to the first dose of investigational product or plan to receive major surgery during the study with exception of the surgical procedures to establish vascular access, biopsy through mediastinoscopy or thoracoscopy; (3) Use of a potent CYP3A4 inhibitor within 7 days prior to the first dose of investigational product or a potent CYP3A4 inducer within 21 days prior to the first dose of investigational product; use of the traditional Chinese medicine or traditional Chinese medicine preparation with tumor indication, or traditional Chinese medicine or traditional Chinese medicine preparation with adjuvant anti-tumor effect within two weeks prior to the first dose of investigational product or expected to be required during the study; (4) Having participated in the clinical trial and received the investigational product or device within 4 weeks or at least 5 half-lives prior to the first dose of investigational product; (5) Having received other anti-tumor drugs within 14 days prior to the first dose of investigational product;
* Having a history of other malignant tumor, or other concurrent malignant tumors;
* The toxicity caused by previous anti-tumor therapy has not recovered to <= CTCAE grade 1 (CTCAE 5.0) (except alopecia, sequelae of previous platinum-related neurotoxicity) ;
* Previous interstitial lung disease (ILD), drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy; or having the clinical manifestations of suspected interstitial lung disease;
* Serious gastrointestinal dysfunction, or disease that may affect the intake, transportation or absorption of investigational product;
* Recently active digestive disease
* The patient is prone to bleeding or has active bleeding; Any bleeding event ≥CTCAE grade 3 within 28 days prior to the first study drug;
* Clinically significant prolonged QT interval or other arrhythmia or clinical status considered by investigators that may increase the risk of prolonged QT interval; for example, QTc > 470 ms on ECG at resting state, complete left bundle branch block, degree III atrioventricular block, congenital long QT syndrome, serious hypokalemia, or current use of drugs that may lead to prolonged QT interval;
* Bone marrow reserve, liver, kidney organs and other functions are insufficient;
* There has been an active venous thrombosis event within the last 6 months;
* Known Active hepatitis B virus , hepatitis C virus (positive HCV Ab) or human immunodeficiency virus (positive HIV antibody) infection;
* Infectious disease requiring intravenous medication;
* Known history of mental disease or drug abuse, and currently having an attack or still taking drugs;
* Known or suspected allergy to Furmonertinib or other components of its preparation;
* Female subjects or female partners of male subjects who are pregnant or lactating, or plan to be pregnant during the study;
* Poor compliance, inability to comply with the study procedures, restriction or requirements;
* Other conditions that are considered by investigators as unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Central Nervous System Objective Response Rate (CNS ORR) | Approximately 12 weeks after the last patient begin study treatment
  Proportion of subjects whose CNS tumors are assessed as complete response(CR) or partial response(PR) according to RANO-BM.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 12 weeks after the last patient begin study treatment
  Proportion of subjects whose tumors are assessed as complete response(CR) or partial response(PR) according to RECIST 1.1.
Disease Control Rate (DCR) | Approximately 12 weeks after the last patient begin study treatment
  Proportion of subjects whose tumors are assessed as CR, PR or stable disease (SD) according to RECIST 1.1.
Progression Free Survival (PFS) | Approximately 18 months after the first patient begin study treatment
  The time from the first dose of the study drugs to the progression of the disease or death for any reason according to RECIST 1.1
Overall survival (OS) | Approximately 24 months after the last patient begin study treatment
  The time from the first dose of the study drugs to the death for any reason according to RECIST 1.1
Central Nervous System Disease Control Rate (CNS DCR) | Approximately 12 weeks after the last patient begin study treatment
  Proportion of subjects whose CNS tumors are assessed as CR, PR or stable disease (SD) according to RANO-BM.
Central Nervous System Progression Free Survival (PFS) | Approximately 18 months after the first patient begin study treatment
  The time from the first dose of the study drugs to the progression of the CNS disease or death for any reason according to RECIST 1.1
Adverse Events (AEs) | rom the start of study drug to 28 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0

OTHER OUTCOMES:
Change from baseline and time to deterioration in gene mutation spectrum of ctDNA | Approximately 18 months from the last patient begin study treatment
  Gene mutation spectrum of ctDNA will be detected by NGS. The development of resistance will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yang, Doctor, Principal Investigator — Cancer Hospital, CAMS

IPD SHARING:
Plan to Share IPD: No